CLINICAL TRIAL: NCT04444635
Title: Serratus Anterior Plane Block in Pediatric Patients Undergoing Thoracic Surgeries: A Randomized Controlled Trial
Brief Title: Serratus Anterior Plane Block in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelaziz Ismail, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N110-2020
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Anesthesia, Local
Keywords: Serratus anterior plane block; Pediatric; Thoracotomy
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blindness will be achieved by patient codes which will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A physician not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anaesthesiologist who is expert in doing the serratus anterior plane block in patients included within the block group. This expert anaesthesiologist will not be involved in collecting data but another anaesthesia doctor will be responsible for patient management and collecting the intraoperative and postoperative data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plan block plus fentanyl infusion (Active Comparator): The patients will receive serratus anterior block in addition to continous intraoperative fentanyl infusion.
  Interventions: Procedure: Serratus Anterior Plan Block+ Fentanyl infusion; Drug: Fentanyl
- Fentanyl infusion only (Active Comparator): The patient will receive fentanyl infusion only.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Procedure: Serratus Anterior Plan Block+ Fentanyl infusion — After induction of anesthesia, the patients will be put on the lateral position with the diseased side up. A linear ultrasound transducer will be placed in a sagittal plane over the mid-clavicular region of the thoracic cage.
  Then counting down ribs till the fifth rib will be identified in the mid-axillary line. The following muscles will be identified overlying the fifth rib: the latissimus dorsi (superficial and posterior),teres major (superior) and serratus muscles (deep and inferior). Under complete sterile conditions, the needle (25 G needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus anterior muscle. Then, 2 mg/kg of 0.25% bupivacaine will be injected with continuous ultrasound guidance. In addition to continuous fentanyl infusion
  Other Names: Serratus Anterior Plan Block
  Arms: Serratus Anterior Plan block plus fentanyl infusion
Drug: Fentanyl — Continuous fentanyl infusion throughout the surgical procedure.

SUMMARY:
The aim of this work is to study the efficacy of ultrasound guided serratus anterior plane block in pediatric patients undergoing thoracic surgeries.

It is a randomized controlled trial.

DETAILED DESCRIPTION:
It is a prospective randomized controlled study. It is designed to estimate and compare the analgesic effect of single shot serratus anterior plane block in pediatric patients undergoing thoracic surgeries with fentanyl infusion versus fentanyl infusion alone as the control group. Our primary outcome will be the total dose of intra-operative fentanyl boluses.

Randomization will be achieved by using an online random number generator. Blindness will be achieved by patient codes which will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A physician not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anaesthesiologist who is expert in doing the serratus anterior plane block in patients included within the block group. This expert anaesthesiologist will not be involved in collecting data but another anaesthesia doctor will be responsible for patient management and collecting the intraoperative and postoperative data.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months-3 years.
* American Society of anesthesiology (ASA) I and II.
* Pediatric patients undergoing thoracic surgeries (with anterior thoracotomy incision).

Exclusion Criteria:

* Patients whose parents or legal guardians refusing to participate.
* Preoperative mechanical ventilation.
* Known or suspected coagulopathy.
* Infection at the site of injection.
* Known or suspected allergy to any of the studied drugs.
* Elevated liver enzymes more than the normal values.
* Procedures with anticipated significant hemodynamic stability.
* Renal function impairment (Creatinine value more than 1.2mg/dl or blood urea nitrogen (BUN) more than 20mg/dl).

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
The total dose of postoperative operative fentanyl consumption in the first 24 hours. | 12 months
  The total dose of postoperative operative fentanyl consumption in micrograms in the first 24 hours will be calculated

SECONDARY OUTCOMES:
Total dosage of additional fentanyl boluses usage in micrograms intraoperatively | 12 months
  Total dosage of additional fentanyl boluses usage in micrograms intraoperatively
First rescue analgesia | 12 months
  Time (in minutes) to 1st rescue analgesia (morphine) post operatively which will be defined to be the elapsed time between stoppage of fentanyl infusion and a patient FLACC score equal or more than 4.
Pain assessment postoperatively by Face, Leg, Activity, Cry, Consolability (FLACC) score, minimum is zero, and maximum is 6. | 12 months
  Pain assessment at 30 min, 60 min, 2 hours, 4hours, 8hours postoperatively by FLACC score.
Intra and postoperative heart rate. | 12 months
  Intra and postoperative heart rate.
Intraoperative and postoperative systolic blood pressure. | 12 months
  Intraoperative and postoperative systolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ISMAIL, Lecturer, Study Director — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The patients data are confidential

REFERENCES:
- [Background] Lonnqvist PA, Morton NS. Postoperative analgesia in infants and children. Br J Anaesth. 2005 Jul;95(1):59-68. doi: 10.1093/bja/aei065. Epub 2005 Jan 21. No abstract available. PMID 15668207
- [Background] Senturk M, Ozcan PE, Talu GK, Kiyan E, Camci E, Ozyalcin S, Dilege S, Pembeci K. The effects of three different analgesia techniques on long-term postthoracotomy pain. Anesth Analg. 2002 Jan;94(1):11-5, table of contents. doi: 10.1213/00000539-200201000-00003. PMID 11772793
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Rogers ML, Henderson L, Mahajan RP, Duffy JP. Preliminary findings in the neurophysiological assessment of intercostal nerve injury during thoracotomy. Eur J Cardiothorac Surg. 2002 Feb;21(2):298-301. doi: 10.1016/s1010-7940(01)01104-6. PMID 11825739
- [Result] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989